CLINICAL TRIAL: NCT01001221
Title: A Dose-Escalation, Single Arm, Combination Study of Cabazitaxel With Gemcitabine to Determine The Safety, And Pharmacokinetics In Subjects With Advanced Solid Malignancies
Brief Title: Dose-Escalation, Safety, Pharmacokinetics Study of Cabazitaxel With Gemcitabine In Patients With Solid Tumor
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Maximum tolerated dose not able to be determined
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD11068
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Results first posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Neoplasms, Malignant
MeSH Terms: conditions — Neoplasms | interventions — cabazitaxel; XRP6258; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabazitaxel + gemcitabine (Experimental): Cabazitaxel and gemcitabine on Day 1 then gemcitabine alone on Day 8 every 3 weeks until disease progression or unacceptable toxicities, withdrawal of consent or Investigator's decision.
  On Day 1, cabazitaxel was given either first followed by gemcitabine (part 1a) or after gemcitabine with 1 hour gap between the two infusions (part 1b). Required premedication with antihistamine, corticosteroid and H2 antagonist was administered intravenously 30 minutes before each dose of cabazitaxel.
  Interventions: Drug: cabazitaxel; Drug: gemcitabine

INTERVENTIONS:
Drug: cabazitaxel — Pharmaceutical form: 60 mg/1.5 ml concentrate solution for infusion
  Route of administration: Intravenous infusion over 60 minutes
  Dosage:
  * Study part 1: 15, 20 or 25 mg/m^2 according to pre-defined dose escalation schedule
  * Study part 2: MTD as determined in Study part 1
  Other Names: XRP6258; Jevtana
Drug: gemcitabine — Pharmaceutical form: According to United States Package Insert (USPI)
  Route of administration: Intravenous infusion over 30 minutes
  Dosage:
  * Study part 1: 700, 900 or 1000 mg/m^2 according to pre-defined dose escalation schedule
  * Study part 2: MTD as determined in Study part 1.
  Other Names: Gemzar

SUMMARY:
Primary Objectives:

* Study part 1: To determine the Maximum Tolerated Dose (MTD) and the Dose Limiting Toxicities (DLTs) of cabazitaxel administered as a 1-hour infusion in combination with gemcitabine, every 3 weeks in patients with advanced solid malignancies.
* Study part 2: To determine the antitumor activity of cabazitaxel in combination with gemcitabine, in an additional extended cohort of 15 patients with advanced solid malignancies treated with the defined MTD, as assessed by objective response rate (ORR) according to the revised guideline for Response Evaluation Criteria in Solid Tumours (RECIST 1.1 criteria).

Secondary Objectives:

* To assess the safety profile of the combination regimen of cabazitaxel with gemcitabine.
* To assess the pharmacokinetics (PK) of cabazitaxel, gemcitabine and its metabolite 2',2' difluorodeoxyuridine (dFdU) when given in combination.
* To determine Time to Progression (TTP), Objective Response Rate (ORR), and Duration of Response (DR), in the extended cohort of patients treated at the MTD in Part 2 of the study and the patients who received the MTD in Part 1 component.

For study part 1, dose levels were to be escalated according to predefined dose escalation decision rules. The Maximum Administered Dose (MAD) was reached at the dose level when at least 2 patients developed a DLT during the first 3 weeks of treatment. There was no further dose escalation when this dose was achieved. The MTD was defined as the highest dose at which 0 or 1 of 3 to 6 patients, respectively, experienced DLT during the first 3 weeks of treatment.

DETAILED DESCRIPTION:
The study consisted of a screening phase (maximum length of 21-day), a treatment phase with 21-day treatment cycles and a 30-day follow-up visit after the last dose of study medication.

The cut-off date for study part 1 was when last participant completed the first treatment cycle and the subsequent 30 days follow-up.

The cut off date for study part 2 was when all participants experienced disease progression, unacceptable toxicity, consent withdrawal or the last participant had completed 26 weeks or 6 cycles on study treatment, whichever came first.

Participants could continue to be treated on study as long as they were benefiting from study treatment and had not met study withdrawal criteria. After withdrawal from study treatment, further treatment, if any, was at the discretion of the Investigator.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed advanced solid malignancy that is metastatic or unresectable, and for which standard curative measures do not exist.

Exclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) > or =2
* Anticipation of need for a major surgical procedure or radiation therapy during the study treatment
* Absence of completion of all prior chemotherapy, biological therapy, targeted non-cytotoxic therapy > or = 3 weeks; and radiotherapy > or = 4 weeks prior to registration. For part 2 only, prior treatment with radiotherapy, chemoembolization therapy, or cryotherapy is allowed if these therapies are not directed to the areas of measurable disease being used for the purposes of this protocol. (4 weeks of washout period is required prior to start the treatment in Part 2)
* Concurrent treatment in another clinical trial or with any other cancer therapy or patients planning to receive these treatments during the study
* Other concurrent serious illness or medical condition, including active infection or human immunodeficiency virus (HIV) disease
* History of any other malignancy with the exception of adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri
* Patients without resolution of all clinically significant toxic effects (excluding alopecia) of any prior therapy to grade < or = 1 by National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 3.0 or to within the limits listed in the specific inclusion/exclusion criteria
* Other severe acute or chronic medical or psychiatric condition, or significant laboratory abnormality requiring further investigation that may cause undue risk for the patient's safety, inhibit protocol participation, or interfere with interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study
* Symptomatic brain metastases or leptomeningeal disease. Patients with asymptomatic or stable brain metastases are allowed
* Women of childbearing potential not protected by highly effective contraceptive method of birth control. All patients of childbearing potential that do not have a negative pregnancy test within the 7 days prior to registration
* Patients who are pregnant or breastfeeding
* For part 2, absence of measurable disease as defined by the most current version of the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. For the Part 1 component, patients with non-measurable disease are accepted
* Inadequate bone marrow or liver or renal organ function
* Any condition which is considered a contraindication to gemcitabine in the local labelling
* Prior treatment with cabazitaxel within the last 2 years
* History of severe hypersensitivity grade 3 or 4 to taxanes, Polysorbate-80, or to compounds with similar chemical structures

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- United States (4):
  - Investigational Site Number 840002, Detroit, Michigan
  - Investigational Site Number 840005, Cincinnati, Ohio
  - Investigational Site Number 840004, Philadelphia, Pennsylvania
  - Investigational Site Number 840001, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 4 sites in the United States. Since it was not possible to determine the maximum Tolerated Dose (MTD) in study part 1, no participant was enrolled in study part 2 and the study was stopped.
Pre-assignment Details: At each dose level, there was a 1-week gap between the treatment of the first participant and the next 2 participants to evaluate toxicity.
  Before escalating to the next dose level, at least 3 participants were to be evaluable for the criteria defining dose limiting toxicity (DLT).
Groups:
- Part 1: Cabazitaxel + Gemcitabine Dose Level 0: Cabazitaxel 20 mg/m^2 IV followed by gemcitabine 1000 mg/m^2 IV on Day 1 then, gemcitabine 1000 mg/m^2 IV on Day 8
  21-day treatment cycles until disease progression or unacceptable toxicities, withdrawal of consent or Investigator's decision
- Part 1: Cabazitaxel + Gemcitabine Dose Level -1: Cabazitaxel 15 mg/m^2 IV followed by gemcitabine 900 mg/m^2 IV on Day 1 then, gemcitabine 900 mg/m^2 IV on Day 8
  21-day treatment cycles until disease progression or unacceptable toxicities, withdrawal of consent or Investigator's decision
- Part 1: Cabazitaxel + Gemcitabine Dose Level -2: Cabazitaxel 15 mg/m^2 IV followed by gemcitabine 700 mg/m^2 IV on Day 1 then, gemcitabine 700 mg/m^2 IV on Day 8
  21-day treatment cycles until disease progression or unacceptable toxicities, withdrawal of consent or Investigator's decision
- Part 1: Gemcitabine + Cabazitaxel Dose Level 0: gemcitabine 700 mg/m^2 IV followed by cabazitaxel 15 mg/m^2 IV on Day 1 then, gemcitabine 700 mg/m^2 IV on Day 8
  21-day treatment cycles until disease progression or unacceptable toxicities, withdrawal of consent or Investigator's decision
- Part 2: Cabazitaxel + Gemcitabine MTD: Cabazitaxel IV and gemcitabine IV on Day 1 then, gemcitabine IV on Day 8 at the Maximum Tolerated Dose (MTD) as determined in study part 1
  21-day treatment cycles until disease progression or unacceptable toxicities, withdrawal of consent or Investigator's decision
Period: Overall Study
Arm/Group | Part 1: Cabazitaxel + Gemcitabine Dose Level 0 | Part 1: Cabazitaxel + Gemcitabine Dose Level -1 | Part 1: Cabazitaxel + Gemcitabine Dose Level -2 | Part 1: Gemcitabine + Cabazitaxel Dose Level 0 | Part 2: Cabazitaxel + Gemcitabine MTD
Started | 5 | 5 | 3 | 6 | 0 (Inability to determine the MTD during study part 1)
Treated | 5 | 5 | 2 | 6 | 0
Completed 1st Treatment Cycle | 5 | 5 | 2 | 6 | 0
Completed | 0 (Participants treated until disease progression or unacceptable toxicity.) | 0 (Participants treated until disease progression or unacceptable toxicity.) | 0 (Participants treated until disease progression or unacceptable toxicity.) | 0 (Participants treated until disease progression or unacceptable toxicity.) | 0
Not Completed | 5 | 5 | 3 | 6 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 2 | 0
Not completed — Disease progression | 3 | 2 | 2 | 4 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 0
Not completed — Not treated; protocol exclusion | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Cabazitaxel + Gemcitabine Dose Level 0 | Part 1: Cabazitaxel + Gemcitabine Dose Level -1 | Part 1: Cabazitaxel + Gemcitabine Dose Level -2 | Part 1: Gemcitabine + Cabazitaxel Dose Level 0 | Total
Number analyzed (Participants) | 5 | 5 | 3 | 6 | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 60.8 (6.6) | 59.2 (9.2) | 53.0 (14.8) | 56.3 (16.1) | 57.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 3 | 8
  Male | 3 | 3 | 2 | 3 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Asian/Oriental | 0 | 0 | 1 | 0 | 1
  Black | 0 | 1 | 0 | 0 | 1
  Caucasian/White | 4 | 4 | 2 | 6 | 16
  Other | 1 | 0 | 0 | 0 | 1
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.87 (0.32) | 1.82 (0.21) | 1.98 (0.42) | 1.84 (0.12) | 1.87 (0.24)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG criteria:
  * 0: Fully active
  * 1: Ambulatory, carry out work of a light or sedentary nature
  * 2: Ambulatory, capable of all selfcare
  * 3: Capable of limited selfcare, confined to bed or chair more than 50% of waking hours
  * 4: Completely disabled, no selfcare, totally confined to bed or chair
  * 5: Dead
  participants
    0 | 0 | 2 | 1 | 1 | 4
    1 | 5 | 3 | 2 | 5 | 15
    2 | 0 | 0 | 0 | 0 | 0
Primary Tumor Site [Number; unit: participants]
  Bladder | 0 | 0 | 1 | 1 | 2
  Colon | 0 | 1 | 0 | 0 | 1
  Head/neck | 0 | 1 | 1 | 0 | 2
  Lung | 2 | 1 | 1 | 0 | 4
  Muscle/soft tissue | 0 | 0 | 0 | 1 | 1
  Other | 0 | 1 | 0 | 0 | 1
  Ovaries | 0 | 0 | 0 | 1 | 1
  Pancreas | 1 | 1 | 0 | 1 | 3
  Pelvis | 0 | 0 | 0 | 1 | 1
  Prostate | 2 | 0 | 0 | 0 | 2
  Skin | 0 | 0 | 0 | 1 | 1
Histological Type [Number; unit: participants]
  Adenocarcinoma | 2 | 4 | 0 | 2 | 8
  Squamous cell carcinoma | 0 | 1 | 0 | 0 | 1
  Other | 3 | 0 | 3 | 4 | 10
Stage at Diagnosis [Number; unit: participants] — Cancer staging is on a scale of I-IV with higher numbers indicating an increase in progression of the disease.
  Stage I: cancers are localized to one part of the body. Stage II: cancers are early locally advanced. Stage III: cancers are late locally advanced. Stage IV: cancers have often metastasized, or spread to other organs or throughout the body.
  participants
    Stage I | 0 | 0 | 0 | 0 | 0
    Stage II | 0 | 1 | 0 | 0 | 1
    Stage III | 0 | 3 | 0 | 1 | 4
    Stage IV | 5 | 0 | 0 | 2 | 7
    Unknown | 0 | 1 | 3 | 3 | 7
Number of Organs Involved [Mean (Standard Deviation); unit: organs] | 4.0 (1.6) | 2.6 (0.5) | 3.3 (0.6) | 2.0 (0.6) | 2.9 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Dose Limiting Toxicities During Dose Escalation
Description: Dose Limiting Toxicities (DLTs) were defined as clinical adverse events (AE) or laboratory abnormalities considered drug-related as assessed by the Investigator or Sponsor, and achieving a Common Terminology Criteria for Adverse Events v3.0 (CTCAE) severity rating of severe (3) or life-threatening (4).
Time Frame: Day 1 to Day 21 of the first treatment cycle
Population: DLT population: All participants who completed assessments for DLT evaluation for Cycle 1 and either:
  * received study treatment during Cycle 1 and had DLT or
  * did not have DLT and received a full dose of study treatment (no delay/reduction) during Cycle 1 and did not receive hematopoietic growth factors.
Measure: Number; unit: participants
Groups:
- Cabazitaxel + Gemcitabine Dose Level 0: Cabazitaxel 20 mg/m^2 IV followed by gemcitabine 1000 mg/m^2 IV on Day 1 then, gemcitabine 1000 mg/m^2 IV on Day 8
  21-day treatment cycles until disease progression or unacceptable toxicities, withdrawal of consent or Investigator's decision
- Cabazitaxel + Gemcitabine Dose Level -1: Cabazitaxel 15 mg/m^2 IV followed by gemcitabine 900 mg/m^2 IV on Day 1 then, gemcitabine 900 mg/m^2 IV on Day 8
  21-day treatment cycles until disease progression or unacceptable toxicities, withdrawal of consent or Investigator's decision
- Cabazitaxel + Gemcitabine Dose Level -2: Cabazitaxel 15 mg/m^2 IV followed by gemcitabine 700 mg/m^2 IV on Day 1 then, gemcitabine 700 mg/m^2 IV on Day 8
  21-day treatment cycles until disease progression or unacceptable toxicities, withdrawal of consent or Investigator's decision
- Gemcitabine + Cabazitaxel Dose Level 0: Gemcitabine 700 mg/m^2 IV followed by cabazitaxel 15 mg/m^2 IV on Day 1 then, gemcitabine 700 mg/m^2 IV on Day 8
  21-day treatment cycles until disease progression or unacceptable toxicities, withdrawal of consent or Investigator's decision
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 5 | 2 | 5
participants | 2 | 2 | 2 | 2

2. Secondary Outcome: Time To Progression With MTD
Description: Time to progression (TTP) was defined as the time from first treatment administration to first documentation of RECIST-defined objective tumor progression (>=20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of >=1 new lesion and/or unequivocal progression of existing non-target lesions).
  Median TTP was to be estimated using the Kaplan-Meier method. Due to the inability to determine MTD during the study part 1, the analysis was not performed.
Time Frame: Fron Day 1 up to a maximum of 12 months
Groups:
- Cabazitaxel + Gemcitabine MTD: Cabazitaxel IV and gemcitabine IV on Day 1 then, gemcitabine IV on Day 8 at the maximum tolerated dose as determined in study part 1
  21-day treatment cycles until disease progression or unacceptable toxicities, withdrawal of consent or Investigator's decision
Arm/Group | Cabazitaxel + Gemcitabine MTD
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response With MTD
Description: Duration of Response (DR) was defined as the time from the first documentation of RECIST-defined objective tumor response to the first documentation of RECIST-defined objective tumor progression or death.
  Median DR was to be estimated using the Kaplan-Meier method. Due to the inability to determine MTD during the study part 1, the analysis was not performed.
Time Frame: Fron Day 1 up to a maximum of 12 months
Arm/Group | Cabazitaxel + Gemcitabine MTD
Number analyzed (Participants) | 0

4. Secondary Outcome: Participants With Adverse Events
Description: Summary of participants with adverse events (AEs) according to severity and relationship to study drug as assessed by the investigator. The National Cancer Institute Common Terminology Criteria for Adverse Event (NCI-CTCAE), version 3.0 was used to grade the severity of AE.
  Treatment-emergent adverse events (TEAEs) are AEs that occurred or worsened from start of treatment up to 30 days after treatment ceased.
  NCI CTCAE v.3.0 grade 3 =severe and grade 4= life-threatening or disabling.
Time Frame: from first dose of study medication up to 30 days after the last dose of study medication (maximum follow-up of 68 weeks)
Population: all treated (AT) population: All enrolled participants who received at least 1 part of a dose of study treatment
Measure: Number; unit: participants
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 5 | 5 | 2 | 6
participants
  Any AE | 5 | 5 | 2 | 6
  Any TEAE | 5 | 5 | 2 | 6
  - Drug-related TEAE | 5 | 5 | 2 | 6
  Grade 3-4 TEAE | 5 | 5 | 2 | 6
  - Grade 3-4 drug-related TEAE | 4 | 5 | 2 | 6
  Serious TEAE | 5 | 2 | 2 | 4
  - Drug-related serious TEAE | 3 | 2 | 2 | 3
  AE leading to drug withdrawn | 2 | 2 | 0 | 2
  - Drug-related AE leading to drug withdrawn | 0 | 2 | 0 | 1
  AE leading to death | 1 | 0 | 0 | 0
  AE leading to dose reduction | 3 | 4 | 2 | 4
  AE leading to dose delay | 4 | 2 | 1 | 4

5. Post Hoc Outcome: Participant Best Response as Per the Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1
Description: Participant Best response was assessed by investigator using the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1:
  * Complete response (CR): Disappearance of all target lesions, all non-target lesions, and no new lesion. Any pathological lymph nodes must have had reduction in the short axis to <10 mm:
  * Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesion;
  * Progressive disease (PD): >=20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of >=1 new lesion and/or unequivocal progression of existing non-target lesions;
  * Stable disease (SD): not a CR, PR or PD.
Time Frame: Up to a maximum of 22 cycles (median 4 cycles)
Population: all treated (AT) population: All enrolled participants who received at least 1 part of a dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 5 | 5 | 2 | 6
participants
  Complete response | 0 | 0 | 0 | 0
  Partial response | 1 | 1 | 0 | 1
  Stable disease | 2 | 3 | 0 | 3
  Progressive disease | 1 | 1 | 2 | 2
  Not evaluable | 1 | 0 | 0 | 0

6. Secondary Outcome: Pharmacokinetic of Cabazitaxel on Cycle 1: Maximum Plasma Concentration Observed (Cmax)
Description: Blood samples for cabazitaxel assay were collected during cycle 1 and cabazitaxel plasma concentrations were determined using a validated liquid chromatography with tandem mass spectometry (LC-MS/MS) method with a lower limit of quantification (LLOQ) of 1 ng/mL.
  Pharmacokinetic (PK) parameters were calculated from plasma concentrations using non-compartmental analysis.
Time Frame: before the start of infusion and 5 minutes before the end of infusion, then 5, 15, 30 minutes, 1, 2, 3, 5, 7, 10, 24, 48, 72, 120 and 168 hours after the end of infusion
Population: PK population: All enrolled participants who received at least 1 part of a dose of study treatment and had at least 1 post treatment analyzable PK sample, and with no prohibited concomitant medications
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 5 | 4 | 2 | 6
ng/ml | 123 (43.7) | 150 (80.9) | 273 (21.9) | 118 (43.9)

7. Secondary Outcome: Pharmacokinetic of Cabazitaxel on Cycle 1: Time to Maximum Concentration (Tmax)
Time Frame: as for outcome 6
Population: PK population as previously defined
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 5 | 4 | 2 | 6
hours (hr) | 1.00 [0.92 to 1.05] | 0.94 [0.87 to 0.95] | 0.94 [0.88 to 1.00] | 0.93 [0.92 to 1.03]

8. Secondary Outcome: Pharmacokinetic of Cabazitaxel on Cycle 1: Area Under the Time Concentration Curve From Time 0 To the Real Time Tlast (AUClast)
Description: Area under the plasma concentration versus time curve calculated using the trapezoidal method from time 0 to the last measurable concentration at time t.
Time Frame: as for outcome 6
Population: PK population as previously defined
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 5 | 4 | 2 | 6
ng*hr/ml | 556 (500) | 352 (101) | 344 (114) | 315 (208)

9. Secondary Outcome: Pharmacokinetic of Cabazitaxel on Cycle 1: Area Under the Time Concentration Curve (AUC)
Description: Area under the plasma concentration versus time curve extrapolated to infinity
Time Frame: as for outcome 6
Population: PK population as previously defined. Six participants' assays could not be used for AUC.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 3 | 3 | 2 | 3
ng*hr/ml | 876 (730) | 420 (77.3) | 462 (156) | 306 (50.1)

10. Secondary Outcome: Pharmacokinetic of Cabazitaxel on Cycle 1: Terminal Half-life (t1/2z)
Time Frame: as for outcome 6
Population: PK population as previously defined
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 5 | 4 | 2 | 6
hours (hr) | 92.1 (40.3) | 88.3 (35.1) | 75.6 (27.8) | 70.3 (43.1)

11. Secondary Outcome: Pharmacokinetic of Cabazitaxel on Cycle 1: Total Plasma Clearance (CL)
Time Frame: as for outcome 6
Population: PK population as previously defined. Six participants' assays could not be used for CL.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 3 | 3 | 2 | 3
L/hr | 61.0 (38.4) | 64.3 (16.2) | 59.5 (6.38) | 90.8 (7.15)

12. Secondary Outcome: Pharmacokinetic of Cabazitaxel on Cycle 1: Volume of Distribution at Steady State (Vss)
Time Frame: as for outcome 6
Population: PK population as previously defined. One participant's assay could not be used for Vss.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 5 | 4 | 2 | 5
L | 6780 (3250) | 4980 (818) | 3930 (1170) | 5570 (2100)

13. Secondary Outcome: Pharmacokinetic of Cabazitaxel on Cycle 1: Total Plasma Clearance Normalized to Body Surface Area (CL/BSA)
Time Frame: as for outcome 6
Population: PK population as previously defined. Six participants' assays could not be used for CL/BSA.
Measure: Mean (Standard Deviation); unit: L/hr/m^2
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 3 | 3 | 2 | 3
L/hr/m^2 | 32.4 (18.3) | 36.1 (6.58) | 31.9 (12.6) | 49.6 (8.56)

14. Secondary Outcome: Pharmacokinetic of Cabazitaxel on Cycle 1: Volume of Distribution at Steady State Normalized to Body Surface Area (Vss/BSA)
Time Frame: as for outcome 6
Population: PK population as previously defined. One participant's assays could not be used for Vss/BSA.
Measure: Mean (Standard Deviation); unit: L/m^2
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 5 | 4 | 2 | 5
L/m^2 | 3530 (1650) | 2690 (434) | 1980 (8.83) | 3020 (1130)

15. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 1: Maximum Plasma Concentration Observed (Cmax)
Description: Blood samples for gemcitabine assay were collected on Day 1 of cycle 1 at the following timepoints:
  * Cabazitaxel + Gemcitabine: prior the start of cabazitaxel infusion, immediately before the end of gemcitabine infusion, 15, 30 minutes, 1.5, 3.5 and 22.5 hours after the end of gemcitabine infusion;
  * Gemcitabine + cabazitaxel: prior the start of gemcitabine infusion, immediately before the end of gemcitabine infusion, 15, 30 minutes, 1, 1.5, 2.5, 9 and 23.5 hours after the end of cabazitaxel infusion;
  Gemcitabine plasma concentrations were determined using validated LC-MS/MS methods with a LLOQ of 50 ng/mL.
  PK parameters were calculated from plasma concentrations using non-compartmental analysis.
Time Frame: 7 to 9 timepoints from start of Day 1 infusion up to 24h hours after the end of infusion depending on the sequence of treatment on Day 1
Population: PK population as previously defined.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 4 | 5 | 2 | 5
ng/ml | 14600 (6050) | 35600 (27200) | 11400 (3270) | 19000 (9130)

16. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 1: Time to Maximum Concentration (Tmax)
Time Frame: as for outcome 15
Population: PK population as previously defined
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 4 | 5 | 2 | 5
hours (hr) | 0.49 [0.47 to 0.50] | 0.38 [0.37 to 0.55] | 0.60 [0.53 to 0.67] | 0.42 [0.37 to 0.50]

17. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 1: Area Under the Time Concentration Curve From Time 0 To the Real Time Tlast (AUClast)
Time Frame: as for outcome 15
Population: PK population as previously defined
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 4 | 5 | 2 | 5
ng*hr/ml | 7320 (1650) | 16000 (11100) | 6120 (3350) | 9920 (5290)

18. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 1: Area Under the Time Concentration Curve (AUC)
Time Frame: as for outcome 15
Population: PK population as previously defined. Five participants' assays could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 3 | 1 | 5
ng*hr/ml | 6290 (1440) | 21900 (10800) | 8530 (NA) — Single participant in analysis | 9970 (5310)

19. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 1: Terminal Half-life (t1/2z)
Time Frame: as for outcome 15
Population: PK population as previously defined. Five participants' assays could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 3 | 1 | 5
hours | 0.295 (0.118) | 0.254 (0.0570) | 0.202 (NA) — Single participant in analysis | 0.256 (0.0933)

20. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 1: Total Plasma Clearance (CL)
Time Frame: as for outcome 15
Population: PK population as previously defined. Five participants' assays could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 3 | 1 | 5
L/hr | 313 (120) | 85.1 (40.6) | 123 (NA) — Single participant in analysis | 174 (106)

21. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 1: Volume of Distribution at Steady State (Vss)
Time Frame: as for outcome 15
Population: PK population as previously defined. Five participants' assays could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 3 | 1 | 5
L | 135 (86.2) | 28.9 (30.4) | 47.0 (NA) — Single participant in analysis | 51.6 (28.8)

22. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 1: Total Plasma Clearance Normalized to Body Surface Area (CL/BSA)
Time Frame: as for outcome 15
Population: PK population as previously defined. Five participants' assays could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: L/hr/m^2
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 3 | 1 | 5
L/hr/m^2 | 159 (31.3) | 49.8 (27.0) | 78.4 (NA) — Single participant in analysis | 96.4 (62.8)

23. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 1: Volume of Distribution at Steady State Normalized to Body Surface Area (Vss/BSA)
Time Frame: as for outcome 15
Population: PK population as previously defined. Five participants' assays could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: L/m^2
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 3 | 1 | 5
L/m^2 | 66.5 (31.7) | 17.3 (18.9) | 29.9 (NA) — Single participant in analysis | 28.7 (17.4)

24. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 8: Maximum Plasma Concentration Observed (Cmax)
Description: Blood samples for gemcitabine assay were collected on Day 8 of cycle 1 at the following timepoints:
  * Cabazitaxel + Gemcitabine: prior the start of infusion, immediately before the end of infusion, 15, 30 minutes, 1.5, 3.5 and 22.5 hours after the end of infusion;
  * Gemcitabine + cabazitaxel: prior the start of infusion, immediately before the end of infusion, 15, 30 minutes, 1, 1.5, 2.5, 9 and 23.5 hours after the end of infusion;
  Gemcitabine plasma concentrations were determined using validated LC-MS/MS methods with a LLOQ of 50 ng/mL.
  PK parameters were calculated from plasma concentrations using non-compartmental analysis.
Time Frame: 7 to 9 timepoints from start of Day 8 infusion up to 24h hours after the end of infusion depending on the sequence of treatment on Day 1
Population: PK population as previously defined
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 4 | 0 | 3
ng/ml | 10200 (283) | 34500 (30800) |  | 14100 (12200)

25. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 8: Time to Maximum Concentration (Tmax)
Time Frame: as for outcome 24
Population: PK population as previously defined
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 4 | 0 | 3
hours (hr) | 0.52 [0.52 to 0.52] | 0.45 [0.42 to 0.55] |  | 0.47 [0.40 to 0.48]

26. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 8: Area Under the Time Concentration Curve From Time 0 To the Real Time Tlast (AUClast)
Time Frame: as for outcome 24
Population: PK population as previously defined
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 4 | 0 | 3
ng*hr/ml | 5530 (1150) | 15300 (11900) |  | 7710 (6840)

27. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 8: Terminal Half-life (t1/2z)
Time Frame: as for outcome 24
Population: PK population as previously defined. Two participants' assays could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 1 | 3 | 0 | 3
hours (hr) | 0.222 (NA) — Single participant in analysis | 0.282 (0.0218) |  | 0.317 (0.113)

28. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 8: Area Under the Time Concentration Curve (AUC)
Time Frame: as for outcome 24
Population: PK population as previously defined. Two participants' assays could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 1 | 3 | 0 | 3
ng*hr/ml | 6360 (NA) — Single participant in analysis | 18500 (12300) |  | 7780 (6880)

29. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 8: Total Plasma Clearance (CL)
Time Frame: as for outcome 24
Population: PK population as previously defined. Two participants' assays could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 1 | 3 | 0 | 3
L/hr | 262 (NA) — Single participant in analysis | 110 (55.8) |  | 252 (158)

30. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 8: Volume of Distribution at Steady State (Vss)
Time Frame: as for outcome 24
Population: PK population as previously defined. Two participants' assays could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 1 | 3 | 0 | 3
L | 104 (NA) — Single participant in analysis | 36.2 (19.4) |  | 93.3 (51.7)

31. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 8: Total Plasma Clearance Normalized to Body Surface Area (CL/BSA)
Time Frame: as for outcome 24
Population: PK population as previously defined. Two participants' assays could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: L/hr/m^2
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 1 | 3 | 0 | 3
L/hr/m^2 | 157 (NA) — Single participant in analysis | 62.8 (32.7) |  | 143 (93.3)

32. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1 Day 8: Volume of Distribution at Steady State Normalized to Body Surface Area (Vss/BSA)
Time Frame: as for outcome 24
Population: PK population as previously defined. Two participants' assays could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: L/m^2
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 1 | 3 | 0 | 3
L/m^2 | 62.2 (NA) — Single participant in analysis | 20.6 (11.6) |  | 52.3 (28.6)

33. Secondary Outcome: Pharmacokinetic of 2',2' Difluorodeoxyuridine on Cycle 1 Day 1: Maximum Plasma Concentration Observed (Cmax)
Description: Blood samples collected for gemcitabine assay were used to assay gemcitabine metabolite, 2',2' difluorodeoxyuridine(dFdU).
  2',2' difluorodeoxyuridine plasma concentrations were determined using validated LC-MS/MS methods with a LLOQ of 50 ng/mL.
  PK parameters were calculated from plasma concentrations using non-compartmental analysis.
Time Frame: as for outcome 15
Population: PK population as previously defined
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 5 | 5 | 2 | 5
ng/ml | 32200 (10000) | 32500 (10800) | 25500 (8770) | 21100 (5980)

34. Secondary Outcome: Pharmacokinetic of 2',2' Difluorodeoxyuridine on Cycle 1 Day 1: Time to Maximum Concentration (Tmax)
Time Frame: as for outcome 15
Population: PK population as previously defined
Measure: Median (Full Range); unit: hours
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 5 | 5 | 2 | 5
hours | 0.73 [0.50 to 0.77] | 0.77 [0.47 to 0.83] | 0.65 [0.53 to 0.77] | 0.77 [0.50 to 1.47]

35. Secondary Outcome: Pharmacokinetic of 2',2' Difluorodeoxyuridine on Cycle 1 Day 1: Area Under the Time Concentration Curve From Time 0 To the Real Time Tlast (AUClast)
Time Frame: as for outcome 15
Population: PK population as previously defined
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 5 | 5 | 2 | 5
ng*hr/ml | 227000 (27500) | 235000 (47400) | 167000 (47500) | 168000 (57000)

36. Secondary Outcome: Pharmacokinetic of 2',2' Difluorodeoxyuridine on Cycle 1 Day 1: Terminal Half-life (t1/2z)
Time Frame: as for outcome 15
Population: PK population as previously defined
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 5 | 5 | 2 | 5
hours | 9.07 (2.22) | 9.41 (0.837) | 7.96 (1.87) | 12.1 (5.17)

37. Secondary Outcome: Pharmacokinetic of 2',2' Difluorodeoxyuridine on Cycle 1 Day 1: Area Under the Time Concentration Curve (AUC)
Time Frame: as for outcome 15
Population: PK population as previously defined. Two participants' assays could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 5 | 5 | 2 | 3
ng*hr/ml | 273000 (58100) | 285000 (61200) | 191000 (66900) | 151000 (37700)

38. Secondary Outcome: Pharmacokinetic of 2',2' Difluorodeoxyuridine on Cycle 1 Day 8: Maximum Plasma Concentration Observed (Cmax)
Description: as for outcome 33
Time Frame: as for outcome 24
Population: All enrolled participants who received at least 1 part of a dose of study treatment and had at least 1 post treatment analyzable PK sample and with no prohibited concomitant medications.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 5 | 0 | 3
ng/ml | 27400 (3180) | 34800 (8630) |  | 18700 (4740)

39. Secondary Outcome: Pharmacokinetic of 2',2' Difluorodeoxyuridine on Cycle 1 Day 8: Time to Maximum Concentration (Tmax)
Time Frame: as for outcome 24
Population: PK population as previously defined
Measure: Median (Full Range); unit: hours
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 5 | 0 | 3
hours | 0.69 [0.52 to 0.85] | 0.68 [0.55 to 1.02] |  | 0.72 [0.70 to 1.00]

40. Secondary Outcome: Pharmacokinetic of 2',2' Difluorodeoxyuridine on Cycle 1 Day 8: Area Under the Time Concentration Curve From Time 0 To the Real Time Tlast (AUClast)
Time Frame: as for outcome 24
Population: PK population as previously defined
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 5 | 0 | 3
ng*hr/ml | 216000 (3700) | 287000 (77500) |  | 141000 (26400)

41. Secondary Outcome: Pharmacokinetic of 2',2' Difluorodeoxyuridine on Cycle 1 Day 8: Terminal Half-life (t1/2z)
Time Frame: as for outcome 24
Population: PK population as previously defined
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 5 | 0 | 3
hours | 7.29 (1.11) | 8.55 (0.820) |  | 9.10 (0.484)

42. Secondary Outcome: Pharmacokinetic of 2',2' Difluorodeoxyuridine on Cycle 1 Day 8: Area Under the Time Concentration Curve (AUC)
Time Frame: as for outcome 24
Population: PK population as previously defined
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 2 | 5 | 0 | 3
ng*hr/ml | 240000 (11300) | 340000 (100000) |  | 168000 (27600)

43. Secondary Outcome: Pharmacokinetic of Gemcitabine on Cycle 1: Ratio Day 1/Day 8 for AUClast and AUC
Description: Ratio Day 1/Day 8 for AUClast and AUC were calculated to assess the effect of cabazitaxel on gemcitabine exposure.
Time Frame: Day 1 (7 to 9 timepoints from start of infusion up to 24h hours after the end of infusion) and Day 8 (7 to 9 timepoints from start of infusion up to 24h hours after the end of infusion)
Population: Enrolled participants who received at least 1 part of a dose of study treatment and had valid Day 1 and Day 8 PK samples. Valid PK samples included at least 1 post treatment analyzable PK sample and no prohibited concomitant medications.
Measure: Mean (Full Range); unit: ratio
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Number analyzed (Participants) | 1 | 3 | 0 | 3
ratio
  AUClast | 1.15 [NA to NA] — Single participant in analysis | 1.17 [0.661 to 2.49] |  | 1.11 [0.994 to 1.25]
  AUC | 1.15 [NA to NA] — Single participant in analysis | 1.24 [0.660 to 2.47] |  | 1.11 [0.994 to 1.25]

44. Primary Outcome: Objective Response Rate With MTD
Description: Objective response was defined as a confirmed complete response (CR) or a confirmed partial response (PR) during the treatment period, based on RECIST 1.1, as assessed by the Investigator.
  CR: Disappearance of all target lesions, all non-target lesions, and no new lesion. Any pathological lymph nodes must have had reduction in the short axis to <10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesion.
  The objective response rate (ORR) was to be calculated as the proportion of participants with confirmed objective response relative to the total number of participants in the analysis population. Due to the inability to determine MTD during the study part 1, the analysis was not performed.
Time Frame: Fron Day 1 up to a maximum of 12 months
Arm/Group | Cabazitaxel + Gemcitabine MTD
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: from first dose of study medication up to 30 days after the last dose of study medication (maximum follow-up of 68 weeks)
Arm/Group | Cabazitaxel + Gemcitabine Dose Level 0 | Cabazitaxel + Gemcitabine Dose Level -1 | Cabazitaxel + Gemcitabine Dose Level -2 | Gemcitabine + Cabazitaxel Dose Level 0
Serious Adverse Events (participants affected / at risk) | 5/5 | 2/5 | 2/2 | 4/6
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 2/2 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabazitaxel + Gemcitabine Dose Level 0 (N=5) | Cabazitaxel + Gemcitabine Dose Level -1 (N=5) | Cabazitaxel + Gemcitabine Dose Level -2 (N=2) | Gemcitabine + Cabazitaxel Dose Level 0 (N=6)
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Intestinal dilatation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Blood electrolytes abnormal (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabazitaxel + Gemcitabine Dose Level 0 (N=5) | Cabazitaxel + Gemcitabine Dose Level -1 (N=5) | Cabazitaxel + Gemcitabine Dose Level -2 (N=2) | Gemcitabine + Cabazitaxel Dose Level 0 (N=6)
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 1 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 4 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 2 | 2 | 0 | 0
Fatigue (General disorders) | 2 | 4 | 1 | 5
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 1 | 1
Pain (General disorders) | 1 | 0 | 0 | 1
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 1
Generalized oedema (General disorders) | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1
Musosal inflammation (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 3
Pyrexia (General disorders) | 0 | 0 | 1 | 2
Weight decreased (Investigations) | 3 | 1 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
Blood alkalne phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Pharmacokinetic results need to be confirmed due to the limited data available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 45 days in advance of proposed submission, the Investigator should forward a copy of the manuscript or abstract for review by the sponsor, and, if necessary, delay publication or communication for a limited time in order to protect the confidentiality or proprietary nature of any information contained therein.